CLINICAL TRIAL: NCT00536263
Title: An Open-label, Randomized Study of PegIntron in the Treatment of HBeAg Positive Chronic Hepatitis B Patients
Brief Title: PegIntron Treatment of Chronic Hepatitis B e Antigen-Positive Patients (P05170/MK-4031-327)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05170
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG 1.0 mcg/kg weekly (QW) * 24 weeks (Active Comparator): PegIntron 1.0 mcg/kg weekly (QW) * 24 weeks + 24 weeks follow-up
  Interventions: Drug: pegylated interferon alpha-2b
- PEG 1.5 mcg/kg QW * 24 wks (Experimental): PegIntron 1.5 mcg/kg QW * 24 wks + 24 wks follow-up
  Interventions: Drug: pegylated interferon alpha-2b
- PEG 1.5 mcg/kg QW * 48 wks (Experimental): PegIntron 1.5 mcg/kg QW * 48 wks + 24 wks follow-up
  Interventions: Drug: pegylated interferon alpha-2b

INTERVENTIONS:
Drug: pegylated interferon alpha-2b — 1.0 mcg/kg subcutaneously (S.C.) QW for 24 weeks
  Arms: PEG 1.0 mcg/kg weekly (QW) * 24 weeks
Drug: pegylated interferon alpha-2b — 1.5 mcg/kg S.C. QW for 24 weeks
  Arms: PEG 1.5 mcg/kg QW * 24 wks
Drug: pegylated interferon alpha-2b — 1.5 mcg/kg S.C. QW for 48 weeks
  Arms: PEG 1.5 mcg/kg QW * 48 wks

SUMMARY:
The purpose of this study is to determine the efficacy and safety of two dosages of PegIntron for treating hepatitis B e antigen (HBeAg) positive chronic hepatitis B compared with the approved dosage, which is PegIntron 1.0 microgram (mcg)/kg given once a week for 24 weeks. This study compares dosages of (1) 1.5 mcg/kg once a week for 24 weeks and (2) 1.5 mcg/kg once a week for 48 weeks with the approved dosage. All subjects are followed for 24 weeks after their treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic hepatitis B:

  * Serum hepatitis B surface antigen positive for at least 6 months
  * Serum hepatitis B e antigen positive
  * Serum negative for hepatitis B surface and e antibodies
  * Plasma hepatitis B virus deoxyribonucleic acid (DNA) level greater than 20,000 IU/mL
  * Alanine aminotransferase (ALT) 2- to 10-times the upper limit of normal
* Compensated liver disease with certain minimum hematological and serum biochemical criteria

Exclusion Criteria:

* Significant hepatic disease from an etiology other than hepatitis B virus
* Antiviral treatment for hepatitis within previous 6 months
* History of severe psychiatric disease, especially depression
* Unstable or significant cardiovascular disease
* Prolonged exposure to known hepatotoxins such as alcohol or drugs
* Any condition that could interfere with the subject participating in and completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cheng J, Wang Y, Hou J, Luo D, Xie Q, Ning Q, Ren H, Ding H, Sheng J, Wei L, Chen S, Fan X, Huang W, Pan C, Gao Z, Zhang J, Zhou B, Chen G, Wan M, Tang H, Wang G, Yang Y, Mohamed R, Guan R, Lee TH, Chang WH, Zhenfei H, Ye Z, Xu D. Peginterferon alfa-2b in the treatment of Chinese patients with HBeAg-positive chronic hepatitis B: a randomized trial. J Clin Virol. 2014 Dec;61(4):509-16. doi: 10.1016/j.jcv.2014.08.008. Epub 2014 Aug 18. PMID 25200354

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks: PegIntron 1.0 mcg/kg QW * 24 weeks + 24 weeks follow-up
- PEG 1.5 mcg/kg QW * 24 Weeks: PegIntron 1.5 mcg/kg QW * 24 weeks + 24 weeks follow-up
- PEG 1.5 mcg/kg QW * 48 Weeks: PegIntron 1.5 mcg/kg QW * 48 weeks + 24 weeks follow-up
Period: Overall Study
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Started | 225 | 221 | 225 (One (1) participant withdrawn from study for non-compliance.)
Completed | 214 | 207 | 204
Not Completed | 11 | 14 | 21
Not completed — Adverse Event | 5 | 5 | 7
Not completed — Lost to Follow-up | 3 | 4 | 4
Not completed — Subject withdrew - not treatment related | 2 | 0 | 5
Not completed — Subject withdrew - treatment related | 0 | 3 | 2
Not completed — Noncompliance with protocol | 0 | 0 | 1
Not completed — Did not meet protocol eligibility | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- PEG 1.0 mcg/kg QW * 24 Weeks: PegIntron 1.0 mcg/kg QW * 24 weeks + 24 weeks follow-up; treated participants
- PEG 1.5 mcg/kg QW * 24 Weeks: PegIntron 1.5 mcg/kg QW * 24 weeks + 24 weeks follow-up; treated participants
- PEG 1.5 mcg/kg QW * 48 Weeks: PegIntron 1.5 mcg/kg QW * 48 weeks + 24 weeks follow-up; treated participants.
- Total: Total of all reporting groups
Arm/Group | PEG 1.0 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks | Total
Number analyzed (Participants) | 225 | 221 | 224 | 670
Age, Continuous [Mean (Standard Deviation); unit: Years] — Treated Participants
  Years | 28.2 (7.2) | 27.5 (7.1) | 28.4 (7.6) | 28.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated Participants
  Participants
    Female | 54 | 57 | 55 | 166
    Male | 171 | 164 | 169 | 504

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hepatitis B Envelope Antigen (HBe or HBeAg) Loss
Description: HBeAg Loss was tested by Abbott Microparticle Enzyme Immunoassay (MEIA)
Time Frame: 24 weeks after end of treatment (EOT)
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants | 39 | 40 | 70
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; Null hypothesis: no difference in the proportion with HBeAg loss. Based on the targeted sample size, there was 80% statistical power (2-sided 0.05 alpha) to detect a true 36% HBeAg loss rate in this treatment arm versus a true rate of 23% in the control arm; Test type: Superiority or Other; p = 0.860, Cochran-Mantel-Haenszel — P-values are unadjusted; Hochberg's adjustment for multiple comparisons was used to maintain the overall 0.05 significance level in test of superiority using the Cochran-Mantel-Haenszel test; Stratified by genotype; Pairwise rate difference = 0.008, 95% CI 2-sided [-0.063 to 0.079]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by genotype; Pairwise rate difference = 0.139, 95% CI 2-sided [0.061 to 0.217]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; Test type: Non-Inferiority or Equivalence — The noninferiority of PEG 1.5 mcg/kg*24 weeks with respect to PEG 1.5 mcg/kg*48 weeks was to be concluded if the lower bound of the one-sided 95% confidence interval of the difference of the rates (PEG 1.5 mcg/kg*24 weeks minus PEG 1.5 mcg/kg*48 weeks) was greater than the noninferiority margin of -10%; Pairwise rate difference = -0.132, 90% CI 2-sided [-0.198 to -0.065]

2. Secondary Outcome: Number of Participants With HBeAg Loss
Description: HBeAg Loss was tested by assay of Abbott MEIA
Time Frame: Up to Treatment Week 48
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants | 31 | 28 | 43
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; Test type: Superiority or Other; p = 0.700, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = -0.011, 95% CI 2-sided [-0.074 to 0.052]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; Test type: Superiority or Other; p = 0.125, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.054, 95% CI 2-sided [-0.014 to 0.123]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; Test type: Superiority or Other; Pairwise rate difference = -0.065, 90% CI 2-sided [-0.122 to -0.008]

3. Secondary Outcome: HBe Seroconversion
Description: HBe seroconversion was defined as HBeAg Loss and Anti-HBeAg Positive. These were tested by assay of Abbott MEIA.
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 31 | 27 | 40
  24 weeks after EOT | 38 | 36 | 67
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.598, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = -0.016, 95% CI 2-sided [-0.078 to 0.047]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.24, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.041, 95% CI 2-sided [-0.027 to 0.108]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.056, 90% CI 2-sided [-0.112 to -0.001]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.830, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = -0.006, 95% CI 2-sided [-0.075 to 0.063]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.130, 95% CI 2-sided [0.053 to 0.208]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.136, 90% CI [-0.201 to -0.071]

4. Secondary Outcome: Number of Participants With Hepatitis B Virus - Deoxyriboncleic Acid (HBV-DNA) <20,000 IU/mL
Description: HBV-DNA was tested by assay of Roche Cobas Taqman (the test
  lowest limit is 6 IU/mL)
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 46 | 61 | 76
  24 weeks after EOT | 44 | 47 | 75
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.076, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.072, 95% CI 2-sided [-0.007 to 0.151]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.135, 95% CI 2-sided [0.053 to 0.216]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.063, 90% CI 2-sided [-0.135 to 0.009]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.662, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.017, 95% CI 2-sided [-0.058 to 0.092]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.139, 95% CI 2-sided [0.059 to 0.220]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.122, 90% CI 2-sided [-0.191 to -0.053]

5. Secondary Outcome: Number of Participants With HBV-DNA < 200 IU/mL
Description: HBV-DNA was tested by assay of Roche Cobas Taqman (the test lowest limit is 6 IU/mL)
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 10 | 14 | 21
  24 weeks after EOT | 12 | 12 | 22
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.373, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.019, 95% CI 2-sided [-0.023 to 0.061]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.040, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.049, 95% CI 2-sided [0.003 to 0.096]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.030, 90% CI 2-sided [-0.072 to 0.011]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.969, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.001, 95% CI 2-sided [-0.041 to 0.043]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.074, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.045, 95% CI 2-sided [-0.004 to 0.094]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.044, 90% CI 2-sided [-0.085 to -0.003]

6. Secondary Outcome: Number of Participants With HBV-DNA Undetectable
Description: Undetectable HBV-DNA was defined as having a level <6 IU/mL by polymerase chain reaction (PCR).
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 4 | 3 | 8
  24 weeks after EOT | 4 | 3 | 8
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.724, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = -0.004, 95% CI 2-sided [-0.027 to 0.019]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.243, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.018, 95% CI 2-sided [-0.012 to 0.048]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.022, 90% CI 2-sided [-0.046 to 0.002]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.724, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = -0.004, 95% CI 2-sided [-0.027 to 0.019]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.232, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.018, 95% CI 2-sided [-0.012 to 0.048]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.022, 90% CI 2-sided [-0.046 to 0.002]

7. Secondary Outcome: Number of Participants With Biochemical Response
Description: Biochemical response was defined as alanine aminotransferase (ALT) normalization.
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 75 | 86 | 103
  24 weeks after EOT | 63 | 80 | 103
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.219, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.056, 95% CI 2-sided [-0.033 to 0.145]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.126, 95% CI 2-sided [0.037 to 0.216]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.071, 90% CI 2-sided [-0.148 to 0.006]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.067, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.082, 95% CI 2-sided [-0.004 to 0.168]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.180, 95% CI 2-sided [0.092 to 0.268]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.098, 90% CI 2-sided [-0.174 to -0.021]

8. Secondary Outcome: Number of Participants With Combined Response
Description: Combined response was defined as HBV DNA <20,000 IU/mL and HBe seroconversion and alanine aminotransferase (ALT) normalization
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 11 | 11 | 23
  24 weeks after EOT | 18 | 23 | 45
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.995, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.001, 95% CI 2-sided [-0.039 to 0.041]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.031, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.054, 95% CI 2-sided [0.005 to 0.103]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.053, 90% CI 2-sided [-0.094 to -0.012]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.389, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.024, 95% CI 2-sided [-0.030 to 0.078]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.121, 95% CI 2-sided [0.058 to 0.184]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.097, 90% CI 2-sided [-0.152 to -0.041]

9. Secondary Outcome: Hepatitis B Surface Antigen (HBsAg) Loss
Description: HBsAg Loss was tested by assay of Abbott MEIA
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 1 | 1 | 4
  24 weeks after EOT | 1 | 1 | 4
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.991, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.000, 95% CI 2-sided [-0.012 to 0.012]
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.181, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.013, 95% CI 2-sided [-0.006 to 0.033]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.013, 90% CI 2-sided [-0.030 to 0.003]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.971, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.000, 95% CI 2-sided [-0.012 to 0.012]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.179, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.013, 95% CI 2-sided [-0.006 to 0.033]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.013, 90% CI 2-sided [-0.030 to 0.003]

10. Secondary Outcome: Hepatitis B Surface Antigen (HBs) Seroconversion
Description: HBs seroconversion was defined as having HBsAg Loss and Anti-HBs Positive
Time Frame: End of treatment (EOT) and 24 weeks after EOT
Population: Treated participants
Measure: Number; unit: Participants
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 225 | 221 | 224
Participants
  EOT | 0 | 0 | 1
  24 weeks after EOT | 0 | 0 | 2
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; End of treatment; Test type: Superiority or Other; p = 0.991, Cochran-Mantel-Haenszel; Stratified by genotype Due to zero responses in the 2 arms, pairwise rate difference & corresponding 95% confidence interval were not applicable
Statistical Analysis 2: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; p = 0.322, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.004, 95% CI 2-sided [-0.004 to 0.013]
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; End of treatment; Test type: Superiority or Other; Pairwise rate difference = -0.004, 90% CI 2-sided [-0.012 to 0.003]
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.991, Cochran-Mantel-Haenszel; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; p = 0.157, Cochran-Mantel-Haenszel; Stratified by genotype; Pairwise rate difference = 0.009, 95% CI 2-sided [-0.003 to 0.021]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; 24 weeks after EOT; Test type: Superiority or Other; Pairwise rate difference = -0.009, 90% CI 2-sided [-0.019 to 0.001]

11. Secondary Outcome: Change From Baseline in Liver Biopsy Score
Description: Method for biopsy scoring was Knodell Scoring System (Histology Activity Index-HAI Score System):
  Score I (periportal +/- bridging necrosis): 0 (none) to 10 (multilobular necrosis).
  Score II (Intralobular degeneration and focal necrosis): 0 (none) to 4 (Marked [involvement of >2/3 of lobules or nodules]).
  Score III (portal inflammation): 0 (none) to 4 (Marked [dense packing of
  inflammatory cells in >2/3 of portal tracts]).
  Score IV (fibrosis): 0 (none) to 4 (cirrhosis).
Time Frame: Baseline to 24 weeks after end of treatment
Population: Treated participants from designated sites
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks | PEG 1.5 mcg/kg QW * 24 Weeks | PEG 1.5 mcg/kg QW * 48 Weeks
Number analyzed (Participants) | 64 | 64 | 46
Units on a scale
  Baseline | 8.0 (3.06) | 8.4 (2.92) | 8.2 (3.33)
  Change from Baseline | -1.1 (3.57) | -1.7 (3.66) | -1.6 (3.96)
Statistical Analysis 1: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks; Test type: Superiority or Other; p = 0.014, t-test, 2 sided; comparison of post-treatment versus baseline values
Statistical Analysis 2: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; comparison of post-treatment versus baseline values
Statistical Analysis 3: Comparison: PEG 1.5 mcg/kg QW * 48 Weeks; Test type: Superiority or Other; p = 0.010, t-test, 2 sided; comparison of post-treatment versus baseline values
Statistical Analysis 4: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 24 Weeks; Test type: Superiority or Other; p = 0.631, ANCOVA; Treatment group and genotype were the fixed effects and baseline was the covariate; Pairwise rate difference = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 5: Comparison: PEG 1.0 mcg/kg Weekly (QW) * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; Test type: Superiority or Other; p = 0.617, ANCOVA; Treatment group and genotype were the fixed effects and baseline was the covariate; Pairwise rate difference = -0.3, 95% CI 2-sided [-1.4 to 0.8]
Statistical Analysis 6: Comparison: PEG 1.5 mcg/kg QW * 24 Weeks vs PEG 1.5 mcg/kg QW * 48 Weeks; Test type: Superiority or Other; Pairwise rate difference = 0.0, 95% CI 2-sided [-1.1 to 1.1]

ADVERSE EVENTS:
Description: Population was all treated participants.
Arm/Group | PEG 1.0 mcg/kg QW x24 Weeks | PEG 1.5 mcg/kg QW x24 Weeks | PEG 1.5 mcg/kg QW x48 Weeks
Serious Adverse Events (participants affected / at risk) | 10/225 | 11/221 | 15/224
Other Adverse Events (participants affected / at risk) | 173/225 | 169/221 | 182/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG 1.0 mcg/kg QW x24 Weeks (N=225) | PEG 1.5 mcg/kg QW x24 Weeks (N=221) | PEG 1.5 mcg/kg QW x48 Weeks (N=224)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
OCULAR ICTERUS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 3 (4) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 4 (4) | 0 (0) | 1 (1)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
PARATYPHOID FEVER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 4 (4) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 4 (4) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1)
THYROID FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SPEECH DISORDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
MANIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG 1.0 mcg/kg QW x24 Weeks (N=225) | PEG 1.5 mcg/kg QW x24 Weeks (N=221) | PEG 1.5 mcg/kg QW x48 Weeks (N=224)
ASTHENIA (General disorders) | 12 (15) | 25 (40) | 15 (21)
FATIGUE (General disorders) | 35 (106) | 29 (119) | 42 (153)
PYREXIA (General disorders) | 156 (253) | 158 (316) | 168 (444)
WEIGHT DECREASED (Investigations) | 5 (5) | 3 (3) | 16 (19)
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 (9) | 16 (22) | 17 (38)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 (38) | 14 (32) | 12 (53)
MYALGIA (Musculoskeletal and connective tissue disorders) | 54 (108) | 70 (137) | 77 (206)
DIZZINESS (Nervous system disorders) | 18 (37) | 21 (44) | 22 (42)
HEADACHE (Nervous system disorders) | 47 (116) | 66 (187) | 59 (178)
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 (16) | 19 (19) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees not to publish/present any interim results of the study without prior written consent of the sponsor. The PI further agrees to provide 45 days written notice to the sponsor prior to submission for publication/presentation to permit the sponsor to review copies of abstracts/manuscripts which report any study results. The sponsor shall have the right to review and comment. If the parties disagree the PI agrees to meet with the sponsor to discuss and resolve.